CLINICAL TRIAL: NCT03366623
Title: Hospitalized Children's Pain Experience. Effect and Influence of Intervention With the Hospital Clown in Acute and Repeated Painful Procedures. A Mixed Method Study.
Brief Title: Procedural Pain in Children: Intervention With the Hospital Clown
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Principal Investigator, Helle Nygård kristensen, Ph.d. student, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pediatric pain 2017
Record Dates: First submitted 2017-11-30; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Pain, Acute; Venous Puncture; Children, Adult
Keywords: Pain assessment; Self report; Hospital clown intervention
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital clown intervention (Other): The performance of the hospital clown included creating a relation with the child by using different techniques in the venipuncture procedure.
  The hospital clown used distraction techniques with music, songs, toys, fake tattoos (a small sticker/label with a picture applied to the skin with water), dream journeys, storytelling and making agreements in collaboration with the child, parents and healthcare personnel.
  Interventions: Behavioral: Hospital clown
- No hospital clown intervention (Other): The clinical staff, defined as pediatric nurses and biomedical laboratory technologists, assisted the child in the venipuncture procedure with conventional communication, comfort and care techniques.
  Interventions: Behavioral: No hospital clown intervention

INTERVENTIONS:
Behavioral: Hospital clown — Presence of the hospital clown
  Arms: Hospital clown intervention
Behavioral: No hospital clown intervention — Presence of pediatric nurses and biomedical laboratory technologists in the venipuncture procedure.
  Arms: No hospital clown intervention

SUMMARY:
This study evaluates the effect of an intervention with a hospital clown compared to standard care on pain experience for acute hospitalized children receiving venipuncture. Half of the children will receive an intervention with the hospital clown while the other half will receive standard care.

DETAILED DESCRIPTION:
Background: Hospitalized children describe the pain associated with painful procedures as one of the worst experiences during hospitalization. These experiences can be traumatic for children and their families. Most children are acutely hospitalized with no chance to prepare the child for painful procedures, while others experience repeated hospitalizations. Previous negative pain experiences are known to have major consequences for future admissions and procedures. Therefore, there is a need for different interventions for pain relief. In 2004, hospital clowns became a part of the team on pediatric wards in Denmark. International studies have shown positive effects of hospital clowns on preoperative anxiety in children, but there is limited knowledge of the impact on the child's experience related to painful procedures.

The overall purpose of this study is to investigate the effect and impact of the hospital clown as a non-pharmacological intervention on hospitalized children's pain experience and ability to cope during painful procedures in both short and long-term treatment and care.

Methods: A two-faced mixed methods study design with merging and connecting results and findings.

1. A prospective, randomized open-label trial to identify whether exposure to the hospital clown has an effect on pain experience in acute hospitalized children receiving venipuncture.
2. An ethnographic study to uncover the pain experience and ability to cope during painful procedures in short-term hospitalization.
3. An ethnographic study to uncover the influence related to repeated painful procedures, as well as uncover if a relationship may have a potential long-term impact.

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted to the hospital
* Scheduled for the venipuncture procedure
* Not prepared for the procedure before coming to the hospital
* Accompanied by at least one parent

Exclusion Criteria:

* Subjects with developmental disorders who could not cooperate with self- reporting of pain
* Subjects who were unable to speak Danish or English

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-01-18 (Actual)

PRIMARY OUTCOMES:
Pain intensity measure on a FACES Pain Scale combined with a Numerical 0-10 Rating Scale | During a time interval of between 0-5 minutes
  Self-reported pain measure conducted after finishing the venipuncture in the examining room

CONTACTS AND LOCATIONS:
Overall Officials: Helle N Kristensen, Principal Investigator — Aalborg University Hospital

IPD SHARING:
Plan to Share IPD: No